CLINICAL TRIAL: NCT06916208
Title: Study of the Effect of Capsinoid Supplementation on Brown Adipose Tissue in Obese Adolescents
Acronym: ADOBAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Collaborators: Institut Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU_ISP1_2025; 2024-A02660-47 (Other: French National Agency for Drug and Health Product Safety)
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Obese Adolescents; Exercise; Diet Modification; Dietary Supplement
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Adolescents in the control group will receive capsules without active product, but of similar appearance, taste and texture (bought from Ajinomoto® (Ajinomoto Health & Nutrition North America, Inc., Japan) 3 times per day, representing 9mg/day all through the duration of the 4-week multidimensional care program.
  Interventions: Other: Control group (placebo)
- capsinoid supplementation (Experimental): dietary supplementation
  Interventions: Dietary Supplement: capsinoid supplementation

INTERVENTIONS:
Dietary Supplement: capsinoid supplementation — Adolescents in the experimental group will receive active capsules containing dihydrocapsiate (bought from Ajinomoto® (Ajinomoto Health & Nutrition North America, Inc., Japan) 3 times per day, representing 9mg/day all through the duration of the 4-week multidimensional care program.
  Arms: capsinoid supplementation
Other: Control group (placebo) — Regular multidimensional care 4-week program
  Arms: Control group

SUMMARY:
Among the new strategies being considered for the treatment of obesity and its metabolic complications, the activation of brown adipose tissue (BAT) from white adipose tissue looks promising. Interest in the study of BAT has increased over the last 5-10 years in response to the discovery of functional BAT in humans. The BAT is a tissue specialized in regulating energy expenditure by producing heat through the oxidation of fatty acids contained in the multiple lipid droplets of brown adipocytes. This adipose tissue does not play a storage role, but rather an anti-obesogenic one, thanks to its high metabolic and energetic activity.

In addition to exposure to cold, which is the major physiological inducer of brown adipocytes, it seems that exercise and the intake of "adrenergic" foods can activate the TAB and potentially induce a change from white to brown tissue via the production of adrenalin and myokines. Acute and/or chronic effects of thermogenic food supplements have been reported on BAT activation and energy metabolism. The most conclusive of these involve the capsinoids found in sweet peppers and chillies. Weight loss also improves BAT activation.

The BAT has already been identified in children. A decrease in its volume and activity from childhood to adolescence and during puberty has been reported.

The main objective of this randomized controlled double-blind study is to investigate the effects of capsinoid dietary supplementation on BAT activity in obese adolescents.

Our general working hypothesis is that capsinoid supplementation, combined with dietary management, leads to an increase in BAT activity.

ELIGIBILITY:
Inclusion Criteria:

* member or beneficiary of a health insurance scheme
* aged between 11 and 18
* Body Mass Index Z score corresponding to stage 2 obesity according to the curves of Rolland-Cachera et al., 1991 and an absence of weight loss of more than 5% of the total weight over the last 3 months.
* effective contraception (in pubescent females)

Exclusion Criteria:

* known allergy to capsinoids and/or soya
* inflammatory digestive pathology and/or history of digestive tract surgery
* participation in another study or in a period of exclusion determined by a previous study
* pregnant, parturient or breastfeeding
* The holder(s) of parental authority or the adolescent refuse(s) to sign the authorisation or acceptance form, respectively.
* It proves impossible to provide the adolescent or parental guardian(s) with informed information.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Temperature variation between supra-clavicular region and sternal control region pre-post cold stimulus. | at inclusion, and at the end of the 4-week program
  Temperature variation between supra-clavicular region and sternal control region pre-post cold stimulus, in °c. This temperature variation is evaluated using an infrared thermal camera (FLIR) during a cold test.

SECONDARY OUTCOMES:
Changes in cutaneous perfusion | at inclusion, and at the end of the 4-week program
  Cutaneous perfusion is measured in the supra-clavicular region using laser-doppler flowmetry, in PU (perfusion units)
Resting metabolism | at inclusion, and at the end of the 4-week program
  Resting metabolism is measured using indirect calorimetry (ErgoCard CPX and off-line analyses based on Weir equations, in kcal/h and kcal/h/kg
Frequency components of heart rate | at inclusion, and at the end of the 4-week program
  High frequence, Low frequency (and High/low frequency ratio), in ms² and %
Temporal components of heart rate | at inclusion, at the end of the 4-week program
  Time-domain metrics used to assess autonomic nervous system function: SDNN Standard Deviation of NN intervals, in ms; Root Mean Square of Successive Differences, in ms; Percentage of NN50 Intervals, in %
Glycemic profile | at inclusion, at the end of the 4-week program
  glucose concentration, in mmol/ and insulin concentration, in μg/mL, from blood test, combined to calcultate the HOMA-IR, an insulin resistance index as [Fasting Insulin (μg/mL)]*[Fasting Glucose (mmol/L)]/22.5
Lipid profile | at inclusion, at the end of the 4-week program
  triglycerides concentration, in mg/dL; total and HDL cholestérol, mg/dL, from blood test
Catecholamines | at inclusion, and at the end of the 4-week program
  catecholamines concentration from blood, ng/L
brown adipose tissue biomarkers | at inclusion, and at the end of the 4-week program
  irisin, 12-diHOME, 13-diHOME, FG, BMP4, BMP7 concentration from blood test, in ng/L
Anthropometry | at inclusion, and at the end of the 4-week program
  Height, Body mass, in kg and z score, used to calcule the body mass index (BMI, in kg/m2) as body mass/height*height. Fat mass is measured in kg, reported to the body mass in % and to the predicted body surface area to calculate the fat mass index (in kg/m2), body surface area being predicted from the height and body mass.
Eating behavior | at inclusion, and at the end of the 4-week program
  Scores for cognitive restraint, uncontrolled eating and emotional eating from the TFEQ21
Treatment compliance | all through the 4-week program
  The amount of capsules ingested is quantified through a diary filled by nurses in charge of capsules dispensing, and reported in % of the theoretical 3/day
Pubertal development | at inclusion
  Stage of pubertal development using Tanner classification, filled by the medical practioner in charge of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Saint Pierre, Palavas-les-Flots, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osuna-Prieto FJ, Martinez-Tellez B, Sanchez-Delgado G, Aguilera CM, Lozano-Sanchez J, Arraez-Roman D, Segura-Carretero A, Ruiz JR. Activation of Human Brown Adipose Tissue by Capsinoids, Catechins, Ephedrine, and Other Dietary Components: A Systematic Review. Adv Nutr. 2019 Mar 1;10(2):291-302. doi: 10.1093/advances/nmy067. PMID 30624591
- [Background] Martins FF, Martins BC, Teixeira AVS, Ajackson M, Souza-Mello V, Daleprane JB. Brown Adipose Tissue, Batokines, and Bioactive Compounds in Foods: An Update. Mol Nutr Food Res. 2024 Mar;68(6):e2300634. doi: 10.1002/mnfr.202300634. Epub 2024 Feb 25. PMID 38402434
- [Background] Chondronikola M, Beeman SC, Wahl RL. Non-invasive methods for the assessment of brown adipose tissue in humans. J Physiol. 2018 Feb 1;596(3):363-378. doi: 10.1113/JP274255. Epub 2018 Jan 15. PMID 29119565
- [Background] Gilsanz V, Chung SA, Jackson H, Dorey FJ, Hu HH. Functional brown adipose tissue is related to muscle volume in children and adolescents. J Pediatr. 2011 May;158(5):722-6. doi: 10.1016/j.jpeds.2010.11.020. Epub 2010 Dec 18. PMID 21168855
- [Background] Cypess AM, Lehman S, Williams G, Tal I, Rodman D, Goldfine AB, Kuo FC, Palmer EL, Tseng YH, Doria A, Kolodny GM, Kahn CR. Identification and importance of brown adipose tissue in adult humans. N Engl J Med. 2009 Apr 9;360(15):1509-17. doi: 10.1056/NEJMoa0810780. PMID 19357406
- [Background] Chechi K, Nedergaard J, Richard D. Brown adipose tissue as an anti-obesity tissue in humans. Obes Rev. 2014 Feb;15(2):92-106. doi: 10.1111/obr.12116. Epub 2013 Oct 25. PMID 24165204
- See also: opinion of the French National Agency for Food, Environmental and Occupational Health Safety — https://www.anses.fr/fr/content/avis-et-rapports-de-lanses-sur-saisine